CLINICAL TRIAL: NCT01629823
Title: Effect of Positive Airway Pressure on Reducing Airway Reactivity in Patients With Asthma
Brief Title: Effect of Positive Airway Pressure on Reducing Airway Reactivity in Patients With Asthma (CPAP)
Acronym: CPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Lung Association Asthma Clinical Research Centers (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert A. Wise, M.D., Robert A. Wise, M.D, American Lung Association Asthma Clinical Research Centers
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALA-ACRC-13; U01HL108730 (NIH)
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CPAP less than 1 cm H₂O (Sham Comparator)
  Interventions: Device: Continuous Positive Airway Pressure device (Resmed, Swift, Mirage)
- CPAP 10cm H₂O (Experimental)
  Interventions: Device: Continuous Positive Airway Pressure device (Resmed, Swift, Mirage)
- CPAP 5cm H₂O (Experimental)
  Interventions: Device: Continuous Positive Airway Pressure device (Resmed, Swift, Mirage)

INTERVENTIONS:
Device: Continuous Positive Airway Pressure device (Resmed, Swift, Mirage) — Continuous Positive Airway Pressure device (Resmed, Swift, Mirage): Participants will be randomized to one of three pre-set CPAP pressures: less than 1 cm water (H₂O), 5 cm H₂O or 10 cm H₂O. They will be instructed to use the CPAP device every night for 12 weeks. Methacholine airways reactivity will be measured at the end of these 12 weeks and again after a 2-week washout period, 14 weeks after randomization.
  Other Names: ResMed CPAP S9 series: Elite & Escape; Masks: Swift FX, Mirage FX

SUMMARY:
The CPAP trial is a 3-arm parallel design randomized sham-controlled trial. Participants are randomly assigned in equal allocation to one of three treatments: CPAP 10 cm water (H₂O) (high) vs. CPAP 5 cm H₂O (medium) vs. CPAP Sham (less than 1 cm H₂O, Low). The treatment period is 12 weeks with airways reactivity assessed at baseline, 6 and 12 weeks of treatment and after a 2 week washout.

DETAILED DESCRIPTION:
It is now well established that failure to rhythmically apply strain to airway smooth muscle leads to change in the biomechanics of the smooth muscle characterized by shortened resting length and increased sensitivity to pharmacologic constrictors. Patients with asthma have physiologic airway characteristics that recapitulate this condition - increased airway tone and increased sensitivity to methacholine. It is our underlying hypothesis that asthma, although it may be initiated by allergic airway inflammation, is promoted by decreased tidal force fluctuations during recumbent sleep. If this is true, then treatments that increase tidal force fluctuations of airways should reverse these abnormalities. One treatment that increases tidal force fluctuations is continuous positive airway pressure (CPAP). CPAP prevents a fall in end expiratory lung volume and prevents closure of airways in dependent regions of the lung thereby permitting the stresses of tidal breathing to apply strain to airways. Preliminary data in 15 asthmatics showed that 1 week of 10cm H₂O nocturnal CPAP was associated with a remarkable 2.7-fold increase in the concentration of methacholine causing a 20% fall in forced expiratory volume in 1 second (FEV₁) (PC20). The objective of this study is to conduct a randomized, sham-controlled, multicenter study of 5 and 10 cm H₂O CPAP in order to verify these findings; to assess the effect of nocturnal CPAP on airways reactivity; to determine the durability of the effect over 12 weeks; to assess the safety, tolerability and adherence to this treatment; and to explore if there are clinically meaningful benefits. The study will be conducted at 18 centers of the American Lung Association-Asthma Clinical Research Centers (ALA-ACRC) with the Data Coordinating Center (DCC) at Johns Hopkins University.

A substudy of High Resolution Computed Tomography (HRCT) will also be conducted at a subset of the ACRC clinics. A total of 54 subjects (18 per arm)who are randomized in the main study will be voluntarily enrolled in the substudy to compare the structural changes in the airways across treatment groups and to correlate structural changes with the physiological changes. A total of two visits will be conducted. HRCT Visit 1 will be performed after randomization in the main CPAP study, and prior to initiation of CPAP. HRCT Visit 2 will be performed between weeks 10 and 12 of CPAP, at a different day or prior of methacholine challenge testing.Two CT scans will be performed each at different lung volume at each visit (Total of 4 scans for the study duration). The first volume will be at Total Lung Capacity (TLC), followed by another CT scan at Functional Residual Capacity (FRC).

ELIGIBILITY:
Inclusion criteria

* 15 - 60 years of age at V1
* Physician diagnosis of asthma and on prescribed asthma medication for at least the past 12 months at V1
* Pre-bronchodilator FEV₁ greater than or equal to 75% predicted at V1 (to minimize the likelihood that variability in FEV₁ will preclude participants from having methacholine challenges in follow-up visits)
* Airways reactivity: Methacholine bronchial challenge with concentration of methacholine causing a 20% fall in forced expiratory volume in 1 second (PC ₂₀) less than or equal to 8 mg/mL at V1
* Stable asthma defined by no change in treatment, emergency department (ED) visit, hospitalization, or urgent health care visit for asthma for the 8 weeks prior to screening
* Non-smoker for more than 6 months and less than or equal to 10 pack-year history of smoking
* Ability and willingness to provide informed consent
* If receiving immunotherapy, must have had stable therapy for the 8 weeks prior to screening
* Spend a minimum of six hours per night in bed on average
* Willingness to sleep 5 days a week on average in the same place for the next 4 months
* For women of child bearing potential; not pregnant, not lactating and agree to practice and adequate birth control method (abstinence, combination barrier and spermicide, or hormonal) for the duration of the study

Exclusion criteria

* Weight less than or equal to 66 lbs. (30kg) at V1
* BMI greater than or equal to 35 at V1
* Acute respiratory illness in the month prior to screening
* Systemic corticosteroid therapy during the 3 months preceding screening
* History of sleep apnea by self-report High risk of sleep apnea as assessed by Multivariable Apnea Prediction (MAP) Index; high risk defined as probability that is equal to or greater than 20%
* Chronic diseases (other than asthma) that in the opinion of the investigator would interfere with participation in the trial or put the participant at risk by participation, e.g. non-skin cancer, chronic diseases of the lung (other than asthma), chronic heart diseases, endocrine diseases, liver, kidney or nervous system diseases, or immunodeficiency, any pre-existing conditions that may be contraindications to positive airway pressure including: severe bullous lung disease, pneumothorax, pathologically low blood pressure, dehydration, cerebrospinal fluid leak, recent cranial surgery, trauma, bypassed upper (supraglottic) airway
* Known sleep disorders that are currently under treatment by a sleep specialist
* Known intolerance to methacholine
* Absolute contraindications to methacholine that include: current use of beta-adrenergic blocking agent, heart attack or stroke in the last 3 months, uncontrolled hypertension, known aortic aneurysm
* Use of investigative drugs or intervention trials in the 30 days prior to screening or during the duration of the study
* Prior use of CPAP for any reason Homelessness, lack of telephone access, or intention to move within the next 4 months of the trial.
* For blinding purposes, members from the same household cannot participate in the study at the same time.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 209 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Holbrook, PHD, Principal Investigator — Johns Hopkins University
Locations (18):
- United States (18):
  - University of Arizona, Tucson, Arizona
  - University of California, San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami/ University of South Florida, Miami, Florida
  - Illinois Consortium, Chicago, Illinois
  - St. Vincent Hospital and Health Care Center, Inc, Indianapolis, Indiana
  - Louisiana State University Health Sciences Center, The Ernest N. Morial Asthma, Allergy and Respiratory Disease Center, New Orleans, Louisiana
  - University of Missouri, Kansas City School of Medicine, Kansas City, Missouri
  - Washington University/ St. Louis University, St Louis, Missouri
  - Hofstra University School of Medicine, Hempstead, New York
  - Columbia University - New York University Consortium, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center/ Columbus Children's Hospital, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas
  - Northern New England Consortium, Colchester, Vermont
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Holbrook JT, Sugar EA, Brown RH, Drye LT, Irvin CG, Schwartz AR, Tepper RS, Wise RA, Yasin RZ, Busk MF; American Lung Association Airways Clinical Research Centers. Effect of Continuous Positive Airway Pressure on Airway Reactivity in Asthma. A Randomized, Sham-controlled Clinical Trial. Ann Am Thorac Soc. 2016 Nov;13(11):1940-1950. doi: 10.1513/AnnalsATS.201601-043OC. PMID 27398992

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 209 individuals were enrolled in the study. 15 of those participants were excluded from data analysis due to significant data irregularities at one clinical site
Groups:
- CPAP Less Than 1 cm Water (H₂O); CPAP 5cm H₂O; CPAP 10cm H₂O: Continuous Positive Airway Pressure device (Resmed, Swift, Mirage): Participants will be randomized to one of three pre-set CPAP pressures: less than 1 cm water (H₂O), 5 cm H₂O or 10 cm H₂O. They will be instructed to use the CPAP device every night for 12 weeks. Methacholine airways reactivity will be measured at the end of these 12 weeks.
Period: Trial Period
Arm/Group | CPAP Less Than 1 cm Water (H₂O) | CPAP 5cm H₂O | CPAP 10cm H₂O
Started | 66 | 69 | 59
Completed | 53 | 56 | 49
Not Completed | 13 | 13 | 10
Not completed — Missed visit | 11 | 9 | 8
Not completed — Pre-diluent FEV₁ predicted <70% | 1 | 1 | 1
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Out-of-window visit | 0 | 2 | 0
Not completed — Failed to hold medication | 0 | 0 | 1
Period: Washout Period
Arm/Group | CPAP Less Than 1 cm Water (H₂O) | CPAP 5cm H₂O | CPAP 10cm H₂O
Started | 54 | 57 | 50
Completed | 51 | 51 | 50
Not Completed | 3 | 6 | 0
Not completed — Safety | 2 | 5 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CPAP Less Than 1 cm H₂O; CPAP 5cm H₂O; CPAP 10cm H₂O: Continuous Positive Airway Pressure device (Resmed, Swift, Mirage): Participants will be randomized to one of three pre-set CPAP pressures: less than 1 cm water (H₂O), 5 cm H₂O or 10 cm H₂O. They will be instructed to use the CPAP device every night for 12 weeks. Methacholine airways reactivity will be measured at the end of these 12 weeks and again after a 2-week washout period, 14 weeks after randomization.
- Total: Total of all reporting groups
Arm/Group | CPAP Less Than 1 cm H₂O | CPAP 5cm H₂O | CPAP 10cm H₂O | Total
Number analyzed (Participants) | 66 | 69 | 59 | 194
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [23 to 47] | 31 [20 to 40] | 25 [18 to 39] | 31 [20 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 35 | 36 | 113
  Male | 24 | 34 | 23 | 81
Region of Enrollment [Number; unit: participants]
  United States | 66 | 69 | 59 | 194
Asthma Symptom Utility Index (ASUI) Score [Median (Inter-Quartile Range); unit: units on a scale] — The Asthma Symptom Utility Index (ASUI) is a brief, interviewer-administered, patient preference-based scale assessing frequency and severity of selected asthma-related symptoms and treatment side effects. The minimum score is 0 and the maximum score is 1, with lower scores indicating more symptoms.
  units on a scale | 0.89 [0.83 to 0.94] | 0.94 [0.85 to 1.00] | 0.92 [0.86 to 0.98] | 0.92 [0.84 to 0.98]
Asthma Control Test (ACT) Score [Median (Inter-Quartile Range); unit: units on a scale] — The Asthma Control Test (ACT) is a validated self-administered survey utilizing 5 questions to assess asthma control on a scale from 1 (poor control) to 5 (total control) in individuals 12 years and older. By answering all 5 questions a patient with asthma can obtain a score that may range between 5 and 25. Asthma control is considered a good characteristic for a person with asthma and therefore a higher score is considered a better outcome.
  units on a scale | 21 [19 to 23] | 22 [20 to 24] | 22 [20 to 23] | 22 [20 to 23]
Marks Asthma Quality of Life [Median (Inter-Quartile Range); unit: units on a scale] — Marks Asthma Quality of Life Questionnaire (AQLQ) measures physical and emotional asthma specific quality of life during the past four weeks. The minimum score is 0 and the maximum score is 80, with lower scores indicating better quality of life. The scale is for use in adults only (individuals aged 18 or older).
  units on a scale | 9 [5 to 21] | 7 [3 to 11] | 6 [3 to 10] | 7 [4 to 12]
Sinonasal Questionnaire (SNQ-6) [Median (Inter-Quartile Range); unit: units on a scale] — The Sinonasal Questionnaire (SNQ-6) is a six-item questionnaire designed to diagnose chronic sinonasal disease in patients with asthma. This questionnaire asks about runny nose, postnasal drip, need to blow the nose, facial pain or pressure, and nasal obstruction. Possible answers include never (zero points), 1-4 times per month (1 point), 2-6 times per week (2 points), and daily (3 points). The number of points is then averaged. The minimum score is 0 and the maximum score is 3, with higher scores indicating higher frequency of sinonasal disease symptoms.
  units on a scale | 0.8 [0.6 to 1.6] | 0.8 [0.4 to 1.4] | 0.8 [0.4 to 1.2] | 0.8 [0.4 to 1.4]
PC20 [Median (Inter-Quartile Range); unit: mg/mL] — The PC20 is the concentration of methacholine needed to produce a 20% fall in forced expiratory volume in 1 second (FEV₁) from baseline.
  mg/mL | 1.06 [0.47 to 2.95] | 0.96 [0.30 to 2.66] | 0.89 [0.28 to 2.33] | 0.98 [0.33 to 2.74]
FEV₁ [Median (Inter-Quartile Range); unit: L] — FEV₁ stands for forced expiratory volume in one second, the volume that has been exhaled at the end of the first second of forced expiration.
  L | 2.9 [2.4 to 3.5] | 3.1 [2.6 to 3.7] | 3.0 [2.7 to 3.4] | 3.1 [2.6 to 3.6]
Percent-predicted FEV₁ [Median (Inter-Quartile Range); unit: percent] | 90.0 [84.0 to 96.3] | 90.9 [81.9 to 99.9] | 91.8 [80.7 to 98.0] | 90.6 [82.7 to 97.9]
Forced vital capacity (FVC) [Median (Inter-Quartile Range); unit: L] — Forced vital capacity: the determination of the vital capacity from a maximally forced expiratory effort.
  L | 3.9 [3.3 to 4.5] | 4.2 [3.5 to 4.9] | 3.9 [3.4 to 4.5] | 4.1 [3.4 to 4.7]
Daily use of inhaled corticosteroid (ICS) [Number; unit: participants] | 11 | 10 | 10 | 31
Daily use of combined inhaled corticosteroid/long acting beta agonist (ICS/LABA) [Number; unit: participants] | 18 | 23 | 13 | 54
Daily use of anti-leukotriene [Number; unit: participants] | 8 | 9 | 5 | 22
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 25.8 [23.0 to 29.8] | 26.2 [22.3 to 28.9] | 24.1 [22.0 to 28.8] | 25.7 [22.3 to 29.0]
Former smoker [Number; unit: participants] | 12 | 6 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Methacholine Reactivity
Description: The primary outcome measure was the change in provocative concentration of methacholine causing a 20% fall in forced expiratory volume in 1 second (FEV₁) (PC20) from baseline to 12 weeks. Modified American Thoracic Society guidelines were followed for pre-bronchodilator spirometry and methacholine challenge testing using the 5 breath dosimeter technique. Up to eleven doses, each a doubling concentration of methacholine (Provocholine™), were inhaled starting at 0.03 mg/mL until a 20% or greater fall in FEV₁ occurred; the maximum dose was 32 mg/mL. Breaths each of doubling concentrations of methacholine were inhaled from a calibrated DeVilbiss™ 646 nebulizer.
Time Frame: 12 weeks after randomization
Measure: Geometric Mean (95% Confidence Interval); unit: mg/mL
Groups:
- CPAP Less Than 1 cm H2O; CPAP 5cm H2O; CPAP 10cm H2O: Continuous Positive Airway Pressure device (Resmed, Swift, Mirage): Participants will be randomized to one of three pre-set CPAP pressures: less than 1 cm water (H₂O), 5 cm H₂O or 10 cm H₂O. They will be instructed to use the CPAP device every night for 12 weeks. Methacholine airways reactivity will be measured at the end of these 12 weeks and again after a 2-week washout period, 14 weeks after randomization.
Arm/Group | CPAP Less Than 1 cm H2O | CPAP 5cm H2O | CPAP 10cm H2O
Number analyzed (Participants) | 66 | 69 | 59
mg/mL
  PC20, 12-week | 2.13 [1.30 to 3.49] | 1.48 [0.96 to 2.28] | 1.44 [0.91 to 2.27]
  PC20, post-washout (14 weeks) | 1.60 [0.96 to 2.69] | 1.37 [0.91 to 2.07] | 1.27 [0.81 to 2.01]
Statistical Analysis 1: Comparison: CPAP Less Than 1 cm H2O vs CPAP 5cm H2O; Both the 5 and 10cm groups were compared to the control group, <1cm H₂O; Test type: Superiority or Other; p = 0.51, Regression, Linear — Comparison of 5cm group to control. No adjustment for multiple comparisons; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.44 to 1.50]
Statistical Analysis 2: Comparison: CPAP Less Than 1 cm H2O vs CPAP 10cm H2O; Test type: Superiority or Other; p = 0.57, Regression, Linear; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.47 to 1.52]

ADVERSE EVENTS:
Arm/Group | CPAP Less Than 1 cm H₂O | CPAP 5cm H₂O | CPAP 10cm H₂O
Serious Adverse Events (participants affected / at risk) | 1/66 | 1/69 | 0/59
Other Adverse Events (participants affected / at risk) | 34/58 | 35/62 | 25/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP Less Than 1 cm H₂O (N=66) | CPAP 5cm H₂O (N=69) | CPAP 10cm H₂O (N=59)
Ischemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Stroke
Pyleonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) — Kidney infection
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Hospitalization due to chronic blood loss and fatigue
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CPAP Less Than 1 cm H₂O (N=58) | CPAP 5cm H₂O (N=62) | CPAP 10cm H₂O (N=57)
Headache (General disorders) | 15/50 (15) | 11/55 (11) | 14/46 (14)
Increased work breathing (Social circumstances) | 3/55 (3) | 7/60 (7) | 3/56 (3)
Acute upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 7 (7) | 5 (5)
Drying of nose, mouth, and/or throat (General disorders) | 10/55 (10) | 13/59 (13) | 8/55 (8)
Nose irritation (General disorders) | 6/57 (6) | 9/61 (9) | 7/56 (7)
Ear or sinus discomfort (Ear and labyrinth disorders) | 7/57 (7) | 8/60 (8) | 6/56 (6)
Congestion, runny nose, sneezing (General disorders) | 21/52 (21) | 25/52 (25) | 14/46 (14)
Eye irritation (Eye disorders) | 5/56 (5) | 4/61 (4) | 3/51 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No